CLINICAL TRIAL: NCT06209359
Title: Mechanisms of Diuretic Resistance in Heart Failure, Aim 3
Acronym: MsDR Aim 3
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey Testani, Associate Professor of Medicine, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000034404; 1R01DK130997-01 (NIH)
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Diuretic Resistance
Keywords: Diuretic; Cardiomyopathy; Diuretic Resistance
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Ammonium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ammonium chloride (Active Comparator): Participants will be randomized to ammonium chloride vs placebo. On Day 0 and 1, the participant will take ammonium chloride or placebo 75 mmol twice daily.
  On Day 2, the participant will take ammonium chloride 150 mmol or placebo once
  Interventions: Drug: Ammonium Chloride
- Placebo (Placebo Comparator): Participants will be randomized to ammonium chloride vs placebo. On Day 0 and 1, the participant will take ammonium chloride or placebo 75 mmol twice daily.
  On Day 2, the participant will take ammonium chloride 150 mmol or placebo once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ammonium Chloride — Participants will be randomized to receive either ammonium chloride or placebo. Participants will receive randomized drug in combination with IV bumetanide, bendroflumethiazide, and amiloride. Following a washout period, participants will be crossed over to the alternate drug.
  Arms: Ammonium chloride
Drug: Placebo — Participants will be randomized to receive either ammonium chloride or placebo. Participants will receive randomized drug in combination with IV bumetanide, bendroflumethiazide, and amiloride. Following a washout period, participants will be crossed over to the alternate drug.
  Arms: Placebo

SUMMARY:
Randomized double-blind placebo-controlled crossover study design

DETAILED DESCRIPTION:
Briefly, the protocol will begin with pre-study determination of diuretic response at the screening visit via administration of 10 mg IV bumetanide and measuring peak FENa. Participants may proceed to the subsequent study procedures. Participants will begin a study diet provided by the metabolic kitchen five days prior to Day 0. Beginning on day 0, participants will take either NH4Cl or placebo 75mmol twice daily. On day 1, the participant will return to study site and receives the first dose of their twice daily study medication as well as their regular loop diuretic dose given as IV bumetanide, followed by completion of the biospecimen collection protocol and a 24-hour urine collection. On day 2, participants will receive a full 150mmol dose at Hr-2 (75 mmol if pH<7.3-7.25, no NH4Cl if pH<7.25). 2 hours after the IV bumetanide is given, 100mmol of sodium bicarbonate in 750ml of 5% dextrose will be administered to participants that received NH4Cl or 750 ml of lactated Ringer's solution to participants that received placebo (provided blinded by the investigational pharmacy).

After this visit, a washout period will be conducted before the above procedures are repeated with the alternate study medication. The washout period will be a minimum of 10 days and a maximum of 28 days. Five days prior to the end of the washout period, the participant will resume the study diet until the end of the study on day 18. On day 16, the participant will be crossed over to the alternate therapy (NH4Cl or placebo). On day 17, the participant will complete the same procedures as day 1 of the first arm. On day 18, the participant will complete the same procedures as day 2 of the first arm.

The administration of Bendroflumethiazide will occur under a separate ancillary protocol

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure
* No plan for titration/change of heart failure medical or device therapies during the study period.
* Absence of non-elective hospitalizations in the previous 2 months.
* At optimal volume status by symptoms, exam, and dry weight.
* Serum potassium ≤ 5.0 mmol/L
* Serum sodium ≥ 130 milliequivalents/ liter (mEq/L)
* Hemoglobin ≥8 g/dL
* Age >18 years
* Objective evidence of diuretic resistance to a 10mg bumetanide challenge (screening visit may occur under this protocol or HIC2000032328 or HIC2000034315) defined as:

  * FENa <10% and total sodium output <150mmol
  * And at least one of the following criteria:

    * Chronic home furosemide dose greater than or equal to 80mg furosemide equivalents
    * eGFR < 60ml/min
    * Serum chloride <100mmol/L
    * FENa <5% and total sodium output <75mmol on the 2 hour

Exclusion Criteria:

* Glomerular filtration rate (GFR) <20 ml/min/1.73m2
* Use of any non-loop type diuretic in the last 7 days with the exclusion of low dose aldosterone antagonist (e.g., spironolactone ≤50 mg)
* History of flash pulmonary edema or a "brittle" volume sensitive HF phenotype such as amyloid cardiomyopathy
* Hemoglobin < 8 g/dL
* Pregnant or breastfeeding
* Cirrhosis or known liver disease
* History of metabolic or respiratory acidosis within 30 days
* Use of metformin, acetazolamide, or any other agent that could predispose to acidosis
* Patients who are on metformin may be enrolled if their metformin can be safely discontinued for the randomized treatment periods in each arm. Any participants who have consistently elevated blood glucose readings > 200 mg/dL while inpatient will not be enrolled.
* Serum bicarbonate level <24mmol/L at screening visit
* Venous potential of hydrogen(pH) <7.35 at screening visit
* Inability to give written informed consent or comply with study protocol or follow-up visits
* On Lithium therapy
* On pimozide or thioridazine
* Diagnosis of liver failure
* Contraindications or allergy to sulfonamides
* Any contraindication to thiazide diuretic or allergy to thiazide or bendroflumethiazide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of distal sodium reabsorption(ADRNa) between NH4Cl vs. placebo study visits | Day 0 vs Day 1
  Comparison of ADRNa between NH4Cl vs. placebo during study visits using fractional excretion of lithium and fractional excretion of sodium to calculate the ADRNa.
Change in urinary extracellular vesicles (uEV) pendrin/exosomal marker(CD9) with the change in distal sodium reabsorption(ADRNa), compared between the placebo and NH4Cl | Day 2 vs Day 18
  Change in uEV pendrin/CD9 with the change in ADRNa, compared between the placebo and NH4Cl study visits
Change of distal sodium reabsorption(ADRNa) between NH4Cl vs. placebo study visits | Day 2 vs Day 18
  Comparison of ADRNa between NH4Cl vs. placebo during study visits using fractional excretion of lithium and fractional excretion of sodium to calculate the ADRNa.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No